CLINICAL TRIAL: NCT03638141
Title: The Effect of CTLA-4/PD-L1 Blockade Following Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE) in Patients With Intermediate Stage of HCC Using Durvalumab (MEDI4736) and Tremelimumab
Brief Title: CTLA-4 /PD-L1 Blockade Following Transarterial Chemoembolization (DEB-TACE) in Patients With Intermediate Stage of HCC (Hepatocellular Carcinoma) Using Durvalumab and Tremelimumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J18118; IRB00179347 (Other: JHM IRB)
Record Dates: First submitted 2018-08-15; First posted 2018-08-20 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Intermediate Stage of Hepatocellular Carcinoma; Hepatocellular Carcinoma
Keywords: HCC; Durvalumab; Tremelimumab; Immunotherapy; PD-L1; Antibodies; Hepatocellular Carcinoma; CTLA-4; DEB-TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab in combination with Tremelimumab (Experimental): Drug: Durvalumab 1500mg IV + Tremelimumab 300 mg IV , single infusion about 2 weeks after first DEB-TACE procedure.
  Drug: Durvalumab (monotherapy) 1500 mg IV infusion every 4 weeks, for maximum 13 doses/cycles.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500mg IV every 4 weeks for up to a maximum of 13 cycles (about 12 months) or until confirmed disease progression.
  Other Names: MEDI4736
Drug: Tremelimumab — Tremelimumab 300 mg IV in combination with Durvalumab 1500mg about 2 weeks after their first DEB-TACE.
  Other Names: CP-675,206

SUMMARY:
The purpose of this study is to determine the safety and efficacy of immunotherapy durvalumab and tremelimumab combined with DEB-TACE in patients with Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age ≥18 years.
* Patients with diagnosis of HCC either by high-resolution imaging (triple-phase CT or MRI) and/or by tumor biopsy.
* Patient is not on systemic treatment for diagnosis of HCC
* HCC meeting Barcelona Clinic Liver Cancer (BCLC) stage B (intermediate stage), with measurable lesions on CT or MRI and without extrahepatic spread
* Have measurable disease
* Have disease that responds to DEB-TACE
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Child-Pugh Score of A or early B (score ≤8) without clinically significant ascites
* Body weight >30 kg
* Patients must have adequate organ function defined by study-specified laboratory tests.
* Evidence of post-menopausal status or negative pregnancy test
* Willing and able to comply with study procedures
* Willing to undergo a liver biopsy

Exclusion Criteria:

* Anyone involved with the planning and/or conduct of the study.
* Has participated in another investigational study during the last 6 months.
* Any concurrent anticancer therapy or received therapy ≤30 days prior to study.
* Major surgical procedure at the time of study enrollment or within 28 days prior to the first dose of study drug.
* Have a vascular invasion or extrahepatic tumor.
* Main portal vein thrombosis present on imaging.
* Uncontrolled hepatic encephalopathy at time of enrollment. - Ascites within 6 weeks prior to study treatment.
* Any contraindications for embolization.
* Has an active infection such as Tuberculosis, HIV, hepatitis B or C.
* History of another primary malignancy or myeloproliferative disorder.
* History of leptomeningeal carcinomatosis.
* History of active primary immunodeficiency.
* Any unresolved toxicities from previous anticancer therapy.
* Active or prior documented GI bleeding due to ulcer or esophageal varices bleeding within 6 months.
* History or current use of immunosuppressive medications within 14 days prior to study medications.
* Major surgical procedure within 28 days prior to the first dose of IP.
* Has an active known or suspected autoimmune disease.
* Patients with hypothyroidism.
* Any active skin conditions.
* History of allogenic organ transplantation.
* Significant heart disease.
* Patients weighing < 30 kg.
* Patients with celiac disease not controlled by diet alone.
* Patient with uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Have received a live vaccine within 30 days prior to study drug.
* Woman who are pregnant or breastfeeding.
* Known allergy or hypersensitivity to the study drug.
* Have received durvalumab, tremelimumab, anti-PD-1, anti-PD-L1 or anti-CTLA-4 in a prior study.
* Unwilling or unable to follow the study schedule for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana De Jesus-Acosta, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Durvalumab in Combination With Tremelimumab: Drug: Durvalumab 1500mg IV + Tremelimumab 300 mg IV , single infusion about 2 weeks after first DEB-TACE procedure.
  Drug: Durvalumab (monotherapy) 1500 mg IV infusion every 4 weeks, for maximum 13 cycles or until confirmed disease progression.
Period: Overall Study
Arm/Group | Durvalumab in Combination With Tremelimumab
Started (Started = enrolled to study.) | 21
Completed (Completed=received at least one dose of study drug.) | 20
Not Completed | 1
Not completed — 1 subject was removed from the study due to non compliance and was never treated. | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug
Arm/Group | Durvalumab in Combination With Tremelimumab
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Hepatitis B or C [Count of Participants; unit: Participants] — Number of patients who had Hepatitis B or C infection at baseline.
  Participants | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on mRECIST criteria. CR = Disappearance of any intratumoral arterial enhancement in all target lesions, PR = At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions.
Time Frame: up to 26 months
Population: Participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab in Combination With Tremelimumab
Number analyzed (Participants) | 20
Participants | 11

2. Secondary Outcome: Drug-related Toxicity
Description: Number of participants experiencing drug-related adverse events (AE) Grade 3 or higher as defined by CTCAE v5.0
Time Frame: up to 16 months
Population: Participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Durvalumab in Combination With Tremelimumab: Durvalumab 1500mg IV + Tremelimumab 300 mg IV , single infusion about 2 weeks after first DEB-TACE procedure.
  Durvalumab (monotherapy) 1500 mg IV infusion every 4 weeks, for maximum 13 cycles or until confirmed disease progression.
Arm/Group | Durvalumab in Combination With Tremelimumab
Number analyzed (Participants) | 20
Participants
  Any gr 3 or higher AE | 4
  Hepatitis | 1
  Diarrhea | 1
  Myalgia | 1
  Myocarditis | 1
  Myositis | 1
  Nausea | 1
  Pericarditis | 1
  Pruritus | 1
  Rash maculo-papular | 2

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as the time from start of the treatment until the documentation of disease progression according to mRECIST or death due to any cause, whichever occurs first. Estimation based on the Kaplan-Meier curve.
Time Frame: up to 58 months
Population: Participants who received at least one dose of study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab in Combination With Tremelimumab
Number analyzed (Participants) | 20
months | 6.1 [3.3 to NA] — NA Explanation: Upper bound confidence interval was not estimable due to insufficient number of events

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is the time from the start of first dose of study drug to death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Time Frame: up to 58 months
Population: Participants who received at least one dose of study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab in Combination With Tremelimumab
Number analyzed (Participants) | 20
months | 28.8 [15.1 to NA] — NA Explanation: Upper bound confidence interval was not estimable due to insufficient number of events

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 58 months
Description: Participants who received at least one dose of study drug were considered at risk
Groups:
- Durvalumab in Combination With Tremelimumab: Drug: Durvalumab 1500mg IV + Tremelimumab 300 mg IV , single infusion about 2 weeks after first DEB-TACE procedure.
  Drug: Durvalumab (monotherapy) 1500 mg IV infusion every 4 weeks, for maximum 13 doses/cycles.
  Durvalumab: Durvalumab 1500mg IV every 4 weeks for up to a maximum of 13 cycles (about 12 months) or until confirmed disease progression.
  Tremelimumab: Tremelimumab 300 mg IV in combination with Durvalumab 1500mg about 2 weeks after their first DEB-TACE.
Arm/Group | Durvalumab in Combination With Tremelimumab
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 10/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab in Combination With Tremelimumab (N=20)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Autoimmune disorder (hepatitis) (Immune system disorders) | 1 (1)
Post-embolization syndrome (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Multi organ failure (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab in Combination With Tremelimumab (N=20)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 12 (18)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Anal hemorrhage (Gastrointestinal disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 6 (10)
Dizziness (Nervous system disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Dyspnea (Nervous system disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Edema limbs (General disorders) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 16 (24)
Fever (General disorders) | 9 (11)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flu like symptoms (General disorders) | 2 (3)
Gait disturbance (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Pain (biopsy site) (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (7)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (3)
INR increased (Investigations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 (18)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (5)
Weight loss (Investigations) | 7 (11)
White blood cell decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT03638141/Prot_SAP_000.pdf